CLINICAL TRIAL: NCT07273383
Title: Self-sampling for HPV Screening: a Population-based Feasibility Study
Brief Title: Self-sampling for HPV Screening
Acronym: HPVselftest
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jessica Ruel Laliberté, MD Msc, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-5842
Record Dates: First submitted 2025-05-22; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: HPV; Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mail (Experimental): One group will receive and return their self-sampling kit by mail.
  Interventions: Diagnostic Test: HPV self-sampling test
- Community pharmacy (Experimental): A second group will pick up their kit from a community pharmacy and return it by mail.
  Interventions: Diagnostic Test: HPV self-sampling test
- Family planning clinic (Experimental): A third group will collect their kit from a family planning clinic, perform the self-sample on-site, and it will be transported by a local courier network.
  Interventions: Diagnostic Test: HPV self-sampling test
- Vaccination center (Experimental): Finally, a fourth group will retrieve their kit and perform the self-sample at a vaccination center in Sherbrooke, with samples then transported by a local network.
  Interventions: Diagnostic Test: HPV self-sampling test

INTERVENTIONS:
Diagnostic Test: HPV self-sampling test — HPV self-sampling test

SUMMARY:
To offer large-scale HPV self-sampling in Québec, it is essential to first demonstrate the most effective pathway for patient recruitment, proper sample collection, and safe continuity of care.

Hypothesis:

The hypotheses are that HPV self-sampling is a safe and effective screening method that can be implemented in Québec, and that it is a screening method appreciated by patients, reliable, and capable of increasing access to cervical cancer screening - particularly for individuals without a family physician.

Objectives:

The primary objective of this study is to assess the feasibility of a large-scale HPV self-sampling system within the CIUSSS de l'Estrie. Secondary objectives include evaluating the percentage of properly collected samples, the return rate of kits according to the collection method, the HPV positivity rate in a sample of the population based on various risk factors, and finally, assessing patient satisfaction with the self-sampling process and the preferred collection method.

Methodology:

This cross-sectional cohort study will be conducted at the CIUSSS de l'Estrie, CHUS Fleurimont. A total of 1,000 women aged 25-65 will be recruited and divided into four groups of 250 participants each. One group will receive and return their self-sampling kit by mail. A second group will pick up their kit from a community pharmacy and return it by mail. A third group will collect their kit from a family planning clinic, perform the self-sample on-site, and it will be transported by a local courier network. Finally, a fourth group will retrieve their kit and perform the self-sample at a vaccination center in Sherbrooke, with samples then transported by a local network. The specimen will be self-collected using a Copan 552C.80 FLOQ Swab and analyzed with the Cobas HPV test on the Cobas 8800 automated system. All participants will complete a recruitment questionnaire to better characterize the study population and their risk factors. A nurse (Nancy Lapointe) will be responsible for managing the test results. Patients will receive an email 8 to 12 weeks after sending their sample, informing them of their result and the next steps to follow. Four care pathways according to the HPV test result are planned:

1. HPV 16 or 18 positive: Patients will be referred for colposcopy.
2. Positive for HPV other than 16 or 18:Patients will be referred to a nurse-led colposcopy clinic for cervical cytology.
3. HPV negative:Patients will be encouraged to follow Québec's cervical cancer screening recommendations.
4. Inconclusive result: Patients will be advised of the need to repeat cervical cancer screening.

Anticipated Results:

HPV self-sampling is a safe, effective, and reliable screening method that can be implemented in Québec. It is expected to be appreciated by patients and increase access to screening, especially among those without a family physician.

DETAILED DESCRIPTION:
Background:

Over the course of their lifetime, it is estimated that one in 168 women in Canada will be diagnosed with cervical cancer, and one in 478 will die from it. Human Papillomavirus (HPV) is responsible for approximately 99.7% of cervical cancers. Since the 2022 recommendation from INESSS, the Pap test as a primary screening method is being progressively replaced by the HPV test. The acceptability of this test as a primary screening method is already widely endorsed by expert societies, due to its higher sensitivity compared to traditional cytology. In Québec, HPV-based cervical cancer screening is recommended every five years. However, as autonomous self-sampling has not yet been implemented, patients must obtain a prescription, and the sample must be collected by a healthcare professional - a process identical to the administrative pathway of the Pap test. This limits access to screening for patients in remote areas, those without a family physician, those reluctant to undergo a vaginal exam, or those whose busy schedules make it difficult to consult a healthcare provider. Since January 2024, British Columbia has implemented a self-sampling system that can be performed at home. According to a study by Jones et al. (2024), within the first five months post-implementation, 25,154 patients completed a mail-in HPV test, including 4,680 individuals who had never previously been screened. More than 4,000 patients who received and returned their self-sampling HPV test did not have an assigned healthcare provider. Numerous studies on the acceptability and effectiveness of HPV testing have been conducted worldwide. However, very few large-scale feasibility studies have been carried out, and none of this type have been conducted in Québec. In short,

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 25 to 65 years
* Speak and understand French without assistance
* Have a CHUS medical record number
* Have internet access (for completing the forms)
* Have a valid mailing address, email address, and phone number

Exclusion Criteria:

* Known positive HPV status
* History of total hysterectomy
* Inability to provide consent

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Assess the percentage of samples correctly collected by patients (considered compliant) according to the collection method. | 6 weeks after the self-collection kits have been sent
  The primary objective of the study is to assess the feasibility of a large-scale HPV self-sampling system within the CIUSSS de l'Estrie.
Return rate | 6 weeks after the self-collection kits have been sent
  Evaluate the return rate of the kits based on the collection method.

SECONDARY OUTCOMES:
HPV positivity rate | 6 weeks after the self-collection kits have been sent
  Number of patients HPV positive according to different cervical cancer risk factors (smoking, hpv vaccination status)
Patient satisfaction | 6 weeks after the self-collection kits have been sent
  Number of participants who reported being satisfied or very satisfied with the method

CONTACTS AND LOCATIONS:
Locations (1):
- CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No